CLINICAL TRIAL: NCT03555994
Title: An Exploratory Phase 2, Randomised, Double-blind, Placebo-controlled, and Open-label Active Comparator Study to Evaluate the Effect of MEDI0382 on Hepatic Glycogen Metabolism in Overweight and Obese Subjects With Type 2 Diabetes Mellitus.
Brief Title: A Study to Investigate the Effect of MEDI0382 on Hepatic Glycogen Metabolism in Overweight and Obese Subjects With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5670C00022; 2017-005081-22 (EudraCT Number)
Record Dates: First submitted 2018-04-18; First posted 2018-06-14 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: 0382, T2DM, Cotadutide, Overweight, Obese, MEDI0382
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — cotadutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MEDI0382 (Part A) (Experimental): MEDI0382 administered subcutaneously (Part A)
  Interventions: Drug: MEDI0382
- Placebo (Part A) (Placebo Comparator): Placebo comparator administered subcutaneously (Part A)
  Interventions: Drug: Placebo
- Liraglutide (Part B) (Active Comparator): Active comparator administered subcutaneously (Part B)
  Interventions: Drug: Liraglutide
- MEDI0382 (Part B) (Experimental): MEDI0382 administered subcutaneously (Part B)
  Interventions: Drug: MEDI0382
- Placebo (Part B) (Placebo Comparator): Placebo comparator administered subcutaneously (Part B)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI0382 — MEDI0382 administered subcutaneously
  Arms: MEDI0382 (Part A); MEDI0382 (Part B)
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo (Part A); Placebo (Part B)
Drug: Liraglutide — Liraglutide administered subcutaneously
  Arms: Liraglutide (Part B)

SUMMARY:
A phase 2 study in two parts (A & B) designed to evaluate the effect of MEDI0382 on Hepatic Glycogen Metabolism in subjects with Type 2 Diabetes Mellitus (T2DM). Approximately 20 subjects will be enrolled in Part A and approximately 30 subjects in Part B.

DETAILED DESCRIPTION:
This is a 2-part exploratory Phase 2 study.

Part A is a randomised, double-blind, placebo-controlled study to evaluate the effect of MEDI0382 (also known as Cotadutide) administered once daily subcutaneously (SC) for 28 days on hepatic glycogen metabolism in overweight and obese subjects with T2DM. Part A is planned to randomise up to 20 subjects. Subjects from Part A will not be re-enrolled in Part B.

Part B is an exploratory Phase 2 randomised, double-blind, placebo-controlled and open-label active comparator study to evaluate the effect of MEDI0382 on hepatic glycogen metabolism in overweight and obese subjects with T2DM. Part B is planned to randomise approximately 30 subjects (not to exceed a maximum of 35 subjects). Subjects in Part B will be randomised to receive double-blind MEDI0382 or placebo, or open-label liraglutide once daily for 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 27 and ≤ 40 kg/m2 (inclusive) at screening
* Glycated haemoglobin (HbA1c) ≤ 8.0% at screening
* Diagnosed with T2DM with glucose control managed with metformin monotherapy where no significant dose change (increase or decrease ≥ 500 mg/day) has occurred in the 3 months prior to screening

Exclusion criteria:

* Any subject who has received another investigational product as part of a clinical study or a GLP-1 analogue-containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening
* Any subject who has received any of the following medications prior to the start of the study:

  * Herbal preparations or drugs licensed for control of body weight or appetite (eg, orlistat, bupropion naltrexone, phentermine-topiramate, phentermine, lorcaserin)
  * Opiates, domperidone, metoclopramide or other drugs known to alter gastric emptying
  * Glucagon
  * Warfarin
* Any contraindication to magnetic resonance imaging/MRS scanning including claustrophobia or dislike of confined spaces
* Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss), a history of type 1 diabetes mellitus (T1DM) or diabetic ketoacidosis, or if the subject has been treated with daily SC insulin within 90 days prior to screening
* Recurrent unexplained hypoglycaemic episodes (defined as glucose < 3.0 mmol/L or < 54 mg/dL on more than 2 occasions in 6 months prior to screening)
* Significant inflammatory bowel disease, gastroparesis, or other severe disease or surgery affecting the upper GI tract (including weightreducing surgery and procedures) which may affect gastric emptying or could affect the interpretation of safety and tolerability data
* Acute or chronic pancreatitis
* Significant hepatic disease (except for NASH or nonalcoholic fatty liver disease without portal hypertension or cirrhosis) and/or subjects with any of the following results at screening:

  * Aspartate transaminase (AST) ≥ 3 × upper limit of normal (ULN)
  * Alanine transaminase (ALT) ≥ 3 × ULN
  * Total bilirubin ≥ 2 × ULN
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) < 30 mL/minute/1.73m2 at screening (glomerular filtration rate estimated according to Modification of Diet in Renal Disease (MDRD) using MDRD Study Equation IDMS-traceable (International System of Units [SI] units)
* Poorly controlled hypertension defined as:

  * Systolic blood pressure (BP) > 180 mm Hg
  * Diastolic BP > 105 mm Hg After 10 minutes of supine rest and confirmed by repeated measurement at screening.
* Unstable angina pectoris, myocardial infarction, transient ischemic attack or stroke within 3 months prior to screening, or subjects who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening
* Severe congestive heart failure (New York Heart Association Class III or IV)
* Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia
* History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer
* Any positive results for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) antibody
* Substance dependence or history of alcohol abuse and/or excess alcohol intake (defined as > 21 units per week for a male subject, and >14 units per week for a female subject). Subjects must have a negative alcohol test result at screening and prior to randomisation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Folke Sjöberg, MD, Principal Investigator — CTC Clinical Trial Consultants AB; MacDonald, Principal Investigator — Nottingham; Schrauwen, Principal Investigator — Maastricht
Locations (3):
- Research Site, Maastricht, Netherlands
- Research Site, Uppsala, Sweden
- Research Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Parker VER, Robertson D, Erazo-Tapia E, Havekes B, Phielix E, de Ligt M, Roumans KHM, Mevenkamp J, Sjoberg F, Schrauwen-Hinderling VB, Johansson E, Chang YT, Esterline R, Smith K, Wilkinson DJ, Hansen L, Johansson L, Ambery P, Jermutus L, Schrauwen P. Cotadutide promotes glycogenolysis in people with overweight or obesity diagnosed with type 2 diabetes. Nat Metab. 2023 Dec;5(12):2086-2093. doi: 10.1038/s42255-023-00938-0. Epub 2023 Dec 8. PMID 38066113
- See also: d5670C00022-amendment-6_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00022&attachmentIdentifier=14b052c7-03a1-4610-bce7-18d656107496&fileName=d5670C00022-amendment-6_Redacted_TO.pdf&versionIdentifier=
- See also: d5670c00022-sap-ed-3_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00022&attachmentIdentifier=0fe07aa7-0574-44f5-b623-69bd532afade&fileName=d5670c00022-sap-ed-3_Redacted_TO.pdf&versionIdentifier=
- See also: D5670C0022 Study Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00022&attachmentIdentifier=3b205a93-0ee5-49e8-b8b0-aaa25e2424e8&fileName=D5670C0022_Study_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Part A, a total of 21 participants participated in the study from 31 May 2018 (date first participant enrolled for Part A) to 23 November 2018 (date of last participant last visit for Part A) at one site in Sweden.
  In Part B, a total of 30 participants participated in the study from 17 December 2019 (date first participant enrolled for Part B) to 14 April 2021 (date of last participant last visit for Part B) at 2 sites (one in Sweden and one in the Netherlands).
Groups:
- Placebo (Part A): Placebo administered subcutaneously (Part A)
- Placebo (Part B): Placebo administered subcutaneously (Part B)
Period: Overall Study
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
Started | 9 | 12 | 10 | 9 | 11
Completed | 9 | 10 | 10 | 9 | 11
Not Completed | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B) | Total
Number analyzed (Participants) | 9 | 12 | 10 | 9 | 11 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 69.3 (5.7) | 65.8 (7.3) | 65.2 (9.1) | 61.8 (7.5) | 64.0 (10.7) | 65.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 3 | 2 | 17
  Male | 6 | 7 | 6 | 6 | 9 | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 0 | 0 | 0
  ASIAN | 0 | 0 | 0 | 0 | 0 | 0
  BLACK OR AFRICAN AMERICAN | 0 | 0 | 0 | 0 | 0 | 0
  OTHER | 0 | 0 | 0 | 0 | 0 | 0
  WHITE | 9 | 12 | 10 | 9 | 11 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Glycogen Concentration Adjusted for Liver Volume as Measured by MRS at T = 4 Hours Post Standardised Morning Meal From Baseline (Day -1) to the End of 28 Days of Treatment (Part A Only)
Description: To assess the effect of MEDI0382 on hepatic glycogen levels postprandially versus placebo after 28 days of treatment
Time Frame: Day -1 to Day 28
Measure: Least Squares Mean (90% Confidence Interval); unit: mmol/L
Arm/Group | Placebo (Part A) | MEDI0382 (Part A)
Number analyzed (Participants) | 9 | 10
mmol/L | 5.5 [-47.2 to 58.3] | -100.2 [-150.2 to -50.1]
Statistical Analysis 1: Comparison: Placebo (Part A) vs MEDI0382 (Part A); Test type: Superiority; p = 0.023, ANCOVA; Least square mean difference = -105.7, 90% CI [-178.8 to -32.6]

2. Primary Outcome: Percentage Change in Fasting Hepatic Glycogen Concentration Adjusted for Liver Volume as Measured by MRS at T = 24 Hours Post Standardised Morning Meal From Baseline (Day -1) to the End of 35 Days of Treatment (Day 36) (Part B)
Description: To assess the effect of MEDI0382 on hepatic glycogen levels versus placebo after 35 days (Part B) of treatment
Time Frame: Day -1 to Day 36
Measure: Least Squares Mean (90% Confidence Interval); unit: percent change from baseline
Arm/Group | MEDI0382 (Part B) | Placebo (Part B)
Number analyzed (Participants) | 9 | 11
percent change from baseline | -27.02 [-38.04 to -16.01] | -1.15 [-11.09 to 8.79]
Statistical Analysis 1: Comparison: MEDI0382 (Part B) vs Placebo (Part B); Test type: Superiority; p = 0.008, ANCOVA; Least square mean difference = -25.87, 90% CI [-40.88 to -10.86]

3. Secondary Outcome: Percentage Change in Fasting Hepatic Glycogen Concentration Adjusted for Liver Volume as Measured by MRS at T = 24 Hours Post Standardised Morning Meal From Baseline (Day 1) to the End of 35 Days of Treatment (Day 36, Part B Only)
Description: To assess the effect of MEDI0382 on hepatic glycogen levels versus liraglutide after 35 days of treatment (Part B only)
Time Frame: Fom baseline (Day -1) to Day 35
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage change from baseline
Groups:
- Liraglutide: Active comparator administered subcutaneously
Arm/Group | Liraglutide | MEDI0382
Number analyzed (Participants) | 10 | 9
percentage change from baseline | -5.33 [-13.97 to 3.32] | -27.31 [-36.42 to -18.20]
Statistical Analysis 1: Comparison: Liraglutide vs MEDI0382; Test type: Superiority; p = 0.008, ANCOVA; Least Square Mean difference = -21.99, 90% CI [-34.55 to -9.43]

4. Secondary Outcome: Change of Hepatic Fat Fraction From Baseline as Measured by Magnetic Resonance Imaging (Day -1) to the End of 35 Days of Treatment (Part B Only)
Time Frame: Day -1 to Day 36
Measure: Least Squares Mean (90% Confidence Interval); unit: percent
Arm/Group | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
Number analyzed (Participants) | 10 | 9 | 11
percent | -15.40 [-21.09 to -9.72] | -26.26 [-51.13 to -1.39] | 8.79 [-10.46 to 28.05]
Statistical Analysis 1: Comparison: MEDI0382 (Part B) vs Placebo (Part B); Test type: Superiority; p = 0.070, ANCOVA; Least Square Mean difference = -35.06, 90% CI [-66.54 to -3.58]
Statistical Analysis 2: Comparison: Liraglutide (Part B) vs MEDI0382 (Part B); Test type: Superiority; p = 0.030, ANCOVA; Least Square Mean difference = -11.72, 90% CI [-20.13 to -3.30]

5. Secondary Outcome: Development of ADA
Time Frame: Baseline to (Follow-up Period) 28 days post last dose + (3-month poststudy)
Measure: Count of Participants; unit: Participants
Groups:
- Liraglutide: Active comparator administered subcutaneously (Part B)
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | MEDI0382 (Part B) | Liraglutide | Placebo (Part B)
Number analyzed (Participants) | 9 | 12 | 9 | 10 | 11
Participants
  Baseline ADA result | 0 | 0 | 0 | 0 | 0
  Day 28 ADA result for Part A Day 35 ADA result for Part B | 0 | 1 | 3 | 0 | 0
  Follow-up ADA result | 0 | 0 | 3 | 0 | 0
  Post Study ADA result | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Measures of Safety and Tolerability of Daily SC Doses of MEDI0382 Titrated up to a Dose Level of 300μg (Parts A and B) by Assessment of Number of Participants withTreatment Emergent Adverse Events (TEAEs) as Assessed by CTCAE V4.0
Description: Safety and tolerability of daily SC doses of MEDI0382 by assessment of the following using CTCAE V4.0: The number of Treatment Emergent Adverse events (TEAEs)
Time Frame: Post dosing (Day 1) to final follow-up (28 Days post last dose)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
Number analyzed (Participants) | 9 | 12 | 10 | 9 | 11
Participants
  At least one event | 7 | 11 | 8 | 7 | 6
  At least one IP related event | 5 | 7 | 7 | 7 | 3

7. Secondary Outcome: Measures of Safety and Tolerability of Daily SC Doses of MEDI0382 Titrated up to a Dose Level of 300μg (Parts A and B) by Assessment of Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs) as Assessed by CTCAE V4.0
Description: Safety and tolerability of daily SC doses of MEDI0382 by assessment of the following using CTCAE V4.0: The number of Treatment-Emergent Serious Adverse Events (TESAEs)
Time Frame: Post dosing (Day 1) to final follow-up (28 Days post last dose)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
Number analyzed (Participants) | 9 | 12 | 10 | 9 | 11
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Measures of Safety and Tolerability of Daily SC Doses of MEDI0382 Titrated up to a Dose Level of 300μg (Parts A and B) by Assessment of Changes in Heart Rate and Blood Pressure
Description: Number of subjects with clinically significant changes in heart rate (BPM) or systolic and diastolic blood pressure (mmHg)
Time Frame: Post dosing (Day 1) to final follow-up (28 Days post last dose)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
Number analyzed (Participants) | 9 | 12 | 10 | 9 | 11
Participants | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Measures of Safety and Tolerability of Daily SC Doses of MEDI0382 Titrated up to a Dose Level of 300μg (Parts A and B) by Assessment of Changes in ECG
Description: Number of subjects with an ECG determined to be abnormal and clinically significant
Time Frame: Post dosing (Day 1) to final follow-up (28 Days post last dose)
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
Number analyzed (Participants) | 9 | 12 | 10 | 9 | 11
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Measures of Safety and Tolerability of Daily SC Doses of MEDI0382 Titrated up to a Dose Level of 300μg (Parts A and B) by Assessment of Changes in Haematology and Clinical Chemistry Parameters
Description: Number of subjects with clinically significant changes in in haematology and or clinical chemistry parameters
Time Frame: Post dosing (Day 1) to final follow-up (28 Days post last dose)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
Number analyzed (Participants) | 9 | 12 | 10 | 9 | 11
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Post dosing (Day 1) to final follow-up (28 Days post last dose)
Arm/Group | Placebo (Part A) | MEDI0382 (Part A) | Liraglutide (Part B) | MEDI0382 (Part B) | Placebo (Part B)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/10 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/10 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 7/9 | 11/12 | 8/10 | 7/9 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=9) | MEDI0382 (Part A) (N=12) | Liraglutide (Part B) (N=10) | MEDI0382 (Part B) (N=9) | Placebo (Part B) (N=11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 1 (42) | 5 (98) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (14) | 1 (42) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 6 (6) | 1 (1) | 3 (3) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Food craving (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 5 (5) | 1 (3) | 1 (1) | 1 (2)
Apathy (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Daydreaming (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is more than 60 days but less than or equal to 180 days from the date that the communication is submitted to the sponsor for review. The sponsor can make comments and suggestions where pertinent to the communication and the Sponsor can request for an exceptional additional delay.

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03555994/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT03555994/SAP_001.pdf